CLINICAL TRIAL: NCT02874001
Title: French Validation of an Interview Guide to the Announcement of Cancer: the Psycho Oncology Basic Documentation
Brief Title: French Validation of an Interview Guide to Cancer Announcement : the Psycho Oncology Basic Documentation
Acronym: PO-BADO
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Fondation de France (Other); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: IB-2013-PO BADO
Record Dates: First submitted 2016-08-08; First posted 2016-08-22 (Estimated); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Cancer; With Caregiver Support Time; 18 Years and Over
Keywords: psychology; caregiver support time
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of the PO-BADO in its short and long versions that need a standardized validation process with the inclusion of 450 Patients

DETAILED DESCRIPTION:
In the case of confirmation of the PO- Bado long version, that means for 240 patients a caregiver support time longest 15 minutes than usually suggested, since in 6 items of the Po- Bado usually explored in the caregiver support time, add 6 other additional items provided in the long version. This further time, can be considered as an additional contribution to the free expression.

For the 120 patients seen during the validation of the short version , there is no change in the duration of the caregiver support time.

ELIGIBILITY:
Inclusion Criteria:

* cancer
* having a caregiver support time
* Aged 18 years and over

Exclusion Criteria:

* without known psychiatric history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of cancer and having a caregiver support time
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stadelmaier Nena, PhD, Principal Investigator — Institut Bergonié

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stadelmaier N, Gana K, Saada Y, Duguey-Cachey O, Quintard B. Psychometric Properties of the French Adaptation of the Basic Documentation for Psycho-Oncology (Po-Bado): A Distress Screening Tool. Behav Ther. 2017 Sep;48(5):596-602. doi: 10.1016/j.beth.2016.12.001. Epub 2016 Dec 13. PMID 28711110
- [Background] Stadelmaier N, Duguey-Cachet O, Saada Y, Quintard B. The Basic Documentation for Psycho-Oncology (PO-Bado): an innovative tool to combine screening for psychological distress and patient support at cancer diagnosis. Psychooncology. 2014 Mar;23(3):307-14. doi: 10.1002/pon.3421. Epub 2013 Oct 14. PMID 24123416

RESULTS

PARTICIPANT FLOW:
Groups:
- Cancer Patients: Patientswere recruited from a Comprehensive Regional Cancer Centre in France
Period: Overall Study
Arm/Group | Cancer Patients
Started | 252
Completed | 252
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cancer Patients
Number analyzed (Participants) | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 252

OUTCOME MEASURES:

1. Primary Outcome: Reliability of the Questionnaire in Terms of Internal Consistency
Description: Internal consistency assessed using the Cronbach's alpha coefficient. Cronbach's alpha coefficient is the correlation between responses to a questionnaire.
  Cronbach's alpha can take values between 0 and 1. The internal consistency of a test is greater when the correlation between items is high on average.
Time Frame: 2 weeks after diagnosis
Measure: Number; unit: alpha coefficient
Arm/Group | Cancer Patients
Number analyzed (Participants) | 252
alpha coefficient | 0.87

2. Primary Outcome: Reliability of the Questionnaire in Terms of Interrater Reliability
Description: Questionnaires were were recorded and interpreted by nurses. Inter-rater reliability assessed for each item and for the entire scale, based on the selection of four nurses who will independently rate the recorded content of interviews. The conclusions will be based on intraclass correlation coefficients (ICC).
Time Frame: 2 weeks after diagnosis
Population: To estimate the interrater reliability (IRR), interviews of 40 patients were recorded and interpreted by four nurses.
  IRR was assessed using a two-way random, consistency, average-measures intraclass correlation coefficient to assess the degree that coders were consistent in their ratings for each patient.
Measure: Number (95% Confidence Interval); unit: correlation coefficient (range -1 to 1)
Arm/Group | Cancer Patients
Number analyzed (Participants) | 40
correlation coefficient (range -1 to 1) | 0.71 [0.43 to 0.95]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not collected
Description: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not collected
Groups:
- Cancer Patients: Patients were recruited from a Comprehensive Regional Cancer Centre in France
Arm/Group | Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes